CLINICAL TRIAL: NCT05501704
Title: ETHAN: A Phase II Study Comparing Different Endocrine THerapies for mAle Breast caNcer
Brief Title: ETHAN - ET for Male BC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jose Pablo Leone (Other)
Collaborators: Eli Lilly and Company (Industry); Translational Breast Cancer Research Consortium (TBCRC) (Unknown)
Responsible Party: Sponsor-Investigator, Jose Pablo Leone, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-225
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Male Breast Cancer; Hormone Receptor-positive Breast Cancer; Hormone Receptor Negative Breast Carcinoma
Keywords: Male Breast Cancer; Hormone Receptor-positive Breast Cancer; Hormone Receptor Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male | interventions — Tamoxifen; Anastrozole; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Window Phase Arm A: Tamoxifen (Experimental): Participants will be randomly assigned to receive Tamoxifen 1x daily for 3 weeks (21days).
  Interventions: Drug: Tamoxifen
- Window Phase Arm B: Anastrozole (Experimental): Participants will be randomly assigned to receive Anastrozole 1x daily for 3 weeks (21days).
  Interventions: Drug: Anastrozole
- Window Phase Arm C: Anastrozole + Degarelix (Experimental): Participants will be randomly assigned to receive Anastrozole 1x daily for 3 weeks (21days) and Degarelix on day 1 only.
  Interventions: Drug: Anastrozole; Drug: Degarelix
- Neoadjuvant Phase Arm D: Tamoxifen (Experimental): Participants will be randomly assigned to receive Tamoxifen 1x daily for 4 cycles (4 months); each study cycle is 28 days.
  Interventions: Drug: Tamoxifen
- Neoadjuvant Phase Arm E: Tamoxifen + Abemaciclib (Experimental): Participants will be randomly assigned to receive Tamoxifen 1x daily and Abemaciclib 2x daily for 4 cycles (4 months); each study cycle is 28 days.
  Interventions: Drug: Tamoxifen; Drug: Abemaciclib
- Neoadjuvant Phase Arm F: Anastrozole and Degarelix (Experimental): Participants will be randomly assigned to receive Anastrozole 1x daily and Degarelix on day 1 of each cycle for 4 cycles (4 months); each study cycle is 28 days.
  Interventions: Drug: Anastrozole; Drug: Degarelix
- Neoadjuvant Phase Arm G: Anastrozole + Degarelix + Abemaciclib (Experimental): Participants will be randomly assigned to receive Anastrozole 1x daily, Degarelix on day 1 of each cycle and Abemaciclib 2x daily for 4 cycles (4 months); each study cycle is 28 days.
  Interventions: Drug: Anastrozole; Drug: Degarelix; Drug: Abemaciclib

INTERVENTIONS:
Drug: Tamoxifen — Taken orally
  Other Names: Nolvadex; Soltamox
  Arms: Neoadjuvant Phase Arm D: Tamoxifen; Neoadjuvant Phase Arm E: Tamoxifen + Abemaciclib; Window Phase Arm A: Tamoxifen
Drug: Anastrozole — Taken orally
  Other Names: Arimidex
  Arms: Neoadjuvant Phase Arm F: Anastrozole and Degarelix; Neoadjuvant Phase Arm G: Anastrozole + Degarelix + Abemaciclib; Window Phase Arm B: Anastrozole; Window Phase Arm C: Anastrozole + Degarelix
Drug: Degarelix — Subcutaneous (under the skin) injection
  Arms: Neoadjuvant Phase Arm F: Anastrozole and Degarelix; Neoadjuvant Phase Arm G: Anastrozole + Degarelix + Abemaciclib; Window Phase Arm C: Anastrozole + Degarelix
Drug: Abemaciclib — Taken orally
  Other Names: Verzenio
  Arms: Neoadjuvant Phase Arm E: Tamoxifen + Abemaciclib; Neoadjuvant Phase Arm G: Anastrozole + Degarelix + Abemaciclib

SUMMARY:
This research study is looking to see how well male breast cancer responds to preoperative treatment with endocrine therapy and which endocrine therapy regimen is the most effective treatment for male breast cancer.

The drugs used in this study are:

* Tamoxifen
* Anastrozole
* Degarelix
* Abemaciclib

DETAILED DESCRIPTION:
This is an open-label, multicenter, randomized trial for men with stage I-III hormone receptor-positive (HR+)/HER2-negative breast cancer. The trial will have two phases: A 3-week window phase containing endocrine therapy followed by a 4-month treatment phase where participants are treated with one of four endocrine therapy treatment combinations.

Tamoxifen is the standard of care for the treatment of breast cancer in men. Anastrozole is a standard treatment in women with breast cancer and works more effectively than tamoxifen. This study hopes to learn if anastrozole may also be effective in men. Given that gonadal suppression and CDK 4/6 inhibitors have both improved treatment in women with breast cancer, the study hopes to learn how the addition of Degarelix (gonadal suppression) and Abemaciclib (CDK 4/6 inhibitors) work in comparison to standard of care tamoxifen.

The research study procedures include screening for eligibility and study treatment including laboratory evaluations and quality of life questionnaires.

After completion of treatment, participants will be followed for up to 10 years

It is expected that about 60 men will take part in this research study.

Eli Lilly, a pharmaceutical company, is supporting this research study by providing one of the study drugs. This study is also being supported by Johns Hopkins University on behalf of the Translational Breast Cancer Research Consortium (TBCRC).

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years or older, with diagnosis of invasive breast cancer who have not undergone surgical resection of the primary tumor and axillary nodes.
* Stage I, II, or III per American Joint Committee on Cancer (AJCC) staging 8th edition (112).
* Breast cancer must be hormone receptor-positive and HER2-negative according to definition below assessed by local pathology.

  * Hormone receptor-positive is defined as: positivity for at least one of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PR]) by IHC. ER and PR assays are considered positive if there are > 1% positive tumor nuclei in the samples.
  * HER2-negative is defined per the current American Society of Clinical Oncology/College of American Pathologists Clinical Practice Guideline (113).
* Patients with multifocal or multicentric disease are eligible if the treating investigator has determined the patient should be treated as ER-positive and HER2-negative.
* Bilateral breast cancers are allowed if the treating investigator has determined the patient should be treated as ER-positive and HER2-negative.
* Patients with a history of ipsilateral or contralateral DCIS or LCIS are eligible.
* ECOG performance status ≤ 2.
* Required laboratory values demonstrating adequate organ function:

  * ANC ≥ 1000/mm3
  * Hemoglobin ≥ 8 g/dl
  * Platelets ≥ 50,000/mm3
  * Serum creatinine ≤ 3.0 x ULN (institutional)
  * Total bilirubin ≤ 2.0 x ULN (institutional).
  * AST and ALT ≤ 5.0 x ULN (institutional)
* Men with partners of childbearing potential must be willing to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment and for 6 months after the last dose of study treatment.
* Non-English-speaking patients are eligible but will be exempt from patient-completed questionnaires.
* Willing and able to sign informed consent.
* Willing to undergo breast biopsy after completion of window phase.
* Patient is able to swallow oral medications.

Exclusion Criteria:

* Prior endocrine therapy, chemotherapy, radiation therapy, or investigational therapy for the current breast cancer diagnosis.
* Prior endocrine therapy, systemic therapy, radiation therapy, or investigational therapy for any other malignancy within the past 12 months.
* Diagnosis of inflammatory breast cancer (T4d).
* Other concurrent serious diseases that may interfere with planned treatment, including severe cardiac disease, congestive heart failure (CHF) of New York Heart Association (NYHA) Class III or higher, severe pulmonary conditions/illness, uncontrolled infections.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2036-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Ki-67 | At the end of the 3-week window period.
  Ki-67 will be evaluated by ImmunoHistoChemistry (IHC) following consensus recommendations using imaging analysis methods.
RCB index | At time of surgery.
  RCB will be determined using data from each participating institution pathology department, and will be reviewed by the study team pathologist.

SECONDARY OUTCOMES:
Changes in estradiol levels | Baseline and at the end of the three-week window period
  To evaluate the physiologic endocrine changes that occur as a result of treatment with tamoxifen, anastrozole and anastrozole and degarelix as measured by estradiol levels at baseline and at the end of the three-week window period
Changes in testosterone levels | Baseline and at the end of the three-week window period
  To evaluate the physiologic endocrine changes that occur as a result of treatment with tamoxifen, anastrozole and anastrozole and degarelix as measured by testosterone levels at baseline and at the end of the three-week window period
Preoperative Endocrine Prognostic Index (PEPI) score | At time of surgery
  To evaluate the comparative efficacy of the experimental treatments as measured by PEPI score at surgery.

OTHER OUTCOMES:
Grade 3 or Higher Treatment-Related Toxicity Rate | Up to 6 months
  All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.
Trial enrollment | 3 years
  We will evaluate how many patients we are able to enroll to this trial in a period of 3 years
Trial completion | 3 years
  We will evaluate how many of the enrolled participants successfully complete the study protocol
EORTC QLC-C30 questionnaire | Up to 6 months
  Patient-reported outcomes (PROs) measures will be conducted using the EORTC QLC-C30 questionnaire.
Adapted EORTC BR23 questionnaire | Up to 6 months
  Patient-reported outcomes (PROs) measures will be conducted using the EORTC BR23, adapted by replacing female-specific items with male-specific sexual activity/function items from PR25 (Appendix D of protocol) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Pablo Leone, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu